CLINICAL TRIAL: NCT03712592
Title: Physiological Constraints Associated With Trail Running
Acronym: UT4M2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.096
Record Dates: First submitted 2018-10-10; First posted 2018-10-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Muscle Fatigue
MeSH Terms: interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 160km (Experimental)
  Interventions: Other: Pre and post running evaluations
- 40km (Experimental)
  Interventions: Other: Pre and post running evaluations
- 100km (Experimental)
  Interventions: Other: Pre and post running evaluations
- 4x40km (Experimental)
  Interventions: Other: Pre and post running evaluations

INTERVENTIONS:
Other: Pre and post running evaluations — Each visit will include a series of neuromuscular, cardiovascular, blood glucose and body composition evaluations will be performed. The subjects will provide some information about their muscular pain and their food and water intake.
  Finally, for the study of sleep that only concerns participants in the 4x40 km race, a home sleep registration banner will be given to each participant of the event step by step at the arrival of each stage in order to study sleep the next night as well as 2 nights after the arrival of the last stage.

SUMMARY:
The practice of mountain running or "trail" is in full development in France and elsewhere in the world. This sporting practice associates specific physiological constraints related in particular to the duration of the efforts made (several hours) and to the ground (important elevation, technical ground, average altitude). Some studies have allowed the last 10 years to initiate the exploration of the physiological consequences of this type of practice, especially from a muscular point of view. However, some important questions remain to be clarified such as the impact of these sports events on fatigue and muscle recovery, cardiovascular, energy and water balance disturbances caused, induced sleep changes and the kinetics of recovery of the various parameters. . These elements remain in particular to be studied in very different racing contexts as currently developed by the organizers, namely race in one stage from long to very long distances (40 to 160 km) and race in stages (4 days, 4 x 40 km) as encountered in the Grenoble UT4M race (Ultra Tour des 4 Massifs).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* 18-55 years
* Absence of chronic cardiovascular, respiratory, metabolic or neuromuscular disease
* > 3 years of trail running (at least 1 race> 40 km / year completed and a race> 100 km completed (trail group 160 km)
* Medical certificate of no contraindication to the practice of the trail
* Subjects available in Grenoble before and within 15 days after the race
* Subjects affiliated to a social security scheme
* Subjects able to sign informed consent.

Exclusion Criteria:

* Cardiorespiratory, metabolic and neurological diseases
* Non-Echogenic Subjects
* Subjects with chronic sleep disorders
* Psychiatric pathologies or ATCD of behavioral disorders
* Persons refusing to sign the information sheet and the participation agreement,
* persons under guardianship or not subject to a social security scheme,
* Pregnant woman, parturient, breastfeeding mother
* Person deprived of liberty by judicial or administrative decision,
* Person subject to a legal protection measure, who can not be included in clinical trials.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Quantification of the level of ankle extensors fatigue induced by trail | one month and 12 days
  Pre-post-force decrease in muscle contractility of ankle extensors assessed by neurostimulation
Quantification of the level of knee extensors fatigue induced by trail | one month and 12 days
  Pre-post-force decrease in muscle contractility of knee extensors assessed by neurostimulation
Quantification of the level of ankle extensors fatigue induced by trail | one month and 12 days
  Pre-post-force decrease in muscle contractility of infarction assessed by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Besson T, Rossi J, LE Roux Mallouf T, Marechal M, Doutreleau S, Verges S, Millet GY. Fatigue and Recovery after Single-Stage versus Multistage Ultramarathon Running. Med Sci Sports Exerc. 2020 Aug;52(8):1691-1698. doi: 10.1249/MSS.0000000000002303. PMID 32079919